CLINICAL TRIAL: NCT02678780
Title: Trial to Assess the Efficacy of Lenvatinib in Metastatic Neuroendocrine Tumors. (TALENT STUDY)
Brief Title: Lenvatinib Efficacy in Metastatic Neuroendocrine Tumors
Acronym: TALENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: Eisai Limited (Industry); Experior S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETNE1509; 2015-001467-39 (EudraCT Number)
Record Dates: First submitted 2016-02-01; First posted 2016-02-10 (Estimated); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Patients with advanced/metastatic, histologically confirmed, grade 1/2 (G1/G2) of 2010 WHO (World Health Organization) classification neuroendocrine tumors of the pancreas after progression to a previous targeted agent.
  Treatment: Dosing schedule of 24 mg once a day of Lenvatinib (two 10-mg capsules + one 4-mg capsule)
  Interventions: Drug: Lenvatinib
- Cohort B (Experimental): Patients with advanced/metastatic, histologically confirmed, grade 1/2 (G1/G2) of 2010 WHO (World Health Organization) classification neuroendocrine tumors of gastrointestinal tract after progression to somatostatin analogues Treatment: Dosing schedule of 24 mg once a day of Lenvatinib (two 10-mg capsules + one 4-mg capsule)
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib
  Other Names: LENVIMA™

SUMMARY:
This is a prospective, international, multi-center, open label, stratified, exploratory phase II study evaluating the efficacy and safety of lenvatinib in patients with advanced/metastatic, neuroendocrine tumors of the pancreas after progression to a previous targeted agent (cohort A) or gastrointestinal tract after progression to somatostatin analogues (cohort B).

DETAILED DESCRIPTION:
Trial to assess the efficacy of Lenvatinib in metastatic neuroendocrine tumor. The primary endpoint of the study is overall response rate (ORR) by RECIST v 1.1 upon central radiologic assessment.

Number of patients: 110 patients Estimated duration of subject participation: 24 months

ELIGIBILITY:
INCLUSION CRITERIA

Subjects must meet all of the following criteria to be included in this study:

1. Subjects must have histologically confirmed diagnosis of one of the following advanced/metastatic neuroendocrine tumor types:

   1. WHO Classification G1/G2 (Ki67<20% and mitotic count ≤20 mitoses x 10 HPF) pancreatic neuroendocrine tumor
   2. WHO Classification G1/G2 (Ki67<20% and mitotic count ≤20 mitoses x 10 HPF) gastrointestinal neuroendocrine tumor (including stomach, small intestine and colorectal origins).
2. Subjects must have evidence of measurable disease meeting the following criteria:

   1. At least 1 lesion of ≥ 1.0 cm in the longest diameter for a non-lymph node, or ≥ 1.5 cm in the short-axis diameter for a lymph node, which is serially measurable according to RECIST 1.1 (Appendix I) using computerized tomography/magnetic resonance imaging (CT/MRI). If there is only one target lesion and it is a non-lymph node, it should have a longest diameter of ≥ 1.5 cm.
   2. Lesions that have had external beam radiotherapy (EBRT) or loco-regional therapies such as radiofrequency (RF) ablation or liver embolization must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion.
3. Subjects must show evidence of disease progression by radiologic image techniques within 12 months (an additional month will be allowed to accommodate actual dates of performance of scans, i.e., within ≤ 13 months) prior to signing informed consent, according to RECIST 1.1 (Appendix I)
4. Subjects must meet the following inclusion criterion regarding primary tumor site:

   1. Pancreatic origin: progression after a previous targeted agent (including mTOR inhibitors, such as everolimus or antiangiogenic therapies, such as sunitinib, sorafenib, axitinib, bevacizumab within others). Combination therapies in the same treatment line (such as sorafenib plus bevacizumab, chemotherapy plus antiangiogenic drugs) are considered one treatment line and are allowed to be included in the study. Patients must be treated with only one previous line of targeted agent(s)-based therapy.

      Previous therapy with somatostatin analogues and/or interferon is allowed and is not considered as a previous targeted agent therapy.
   2. Gastrointestinal origin: progression after therapy with antitumoral doses of somatostatin analogs (octreotide LAR 30 mg every 28 days or Lanreotide 120 mg every 28 days) and/or interferon treatment.
5. Only for patients with pancreatic origin neuroendocrine tumors, one previous line with chemotherapy is allowed.
6. Concomitant somatostatin analogues are allowed in both cohorts during the study.
7. Patients with known brain metastases who have completed whole brain radiotherapy, stereotactic radiosurgery or complete surgical resection, will be eligible if they have remained clinically stable, asymptomatic and off of steroids for at least one month.
8. All prior chemotherapy or radiation-related toxicities must have resolved to < Grade 2 (following CTCAE V 4.03 grade levels), except alopecia and infertility.
9. Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 1 (Appendix II).
10. Previous liver locoregional therapies, such as (chemo) embolization, radiofrequency or liver-directed (radio) embolization, or systemic peptide-receptor radionucleotide therapy are allowed if the procedure was performed at least 6 months previous the informed consent form signature.
11. Adequately controlled blood pressure with or without antihypertensive medications, defined as BP < 150/90 mmHg at screening and no change in antihypertensive medications within 1 week prior to the Screening Visit.
12. Adequate renal function defined as calculated creatinine clearance ≥ 30 mL/min per the Cockcroft and Gault formula (Appendix III).
13. Adequate bone marrow function, defined as:

    1. Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 ×103/μL).
    2. Platelets ≥ 100,000/mm3 (≥ 100 × 109/L).
    3. Hemoglobin ≥ 9.0 g/dL.
14. Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) ≤ 1.5. Prophylactic low molecular weight heparin therapy is allowed.
15. Adequate liver function:

    1. Bilirubin ≤ 1.5 × the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia or Gilbert's syndrome.
    2. Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 3 × the ULN (≤ 5 × ULN if subject has liver metastases).
16. Males or females age ≥ 18 years at the time of informed consent.
17. All females must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of beta human chorionic gonadotropin (β-hCG) at the baseline visit (and/or within 72h prior to the first dose of study drug).

    Females of childbearing potential must agree to use a highly effective method of contraception (e.g., total sexual abstinence*, an intrauterine device, a double-barrier method such as condom + spermicide or condom + diaphragm with spermicide or have a vasectomized partner with confirmed azoospermia*) throughout the entire study period and for 30 days after study drug administration. The only subjects who will be exempt from this requirement are postmenopausal women (defined as women who have been amenorrheic for at least 12 consecutive months, in the appropriate age group, without other known or suspected primary cause) or subjects who have been sterilized surgically or who are otherwise proven sterile (i.e., bilateral tubal ligation with surgery at least 1 month prior to dosing, hysterectomy, or bilateral oophorectomy with surgery at least 1 month prior to dosing).

    The women using oral hormonal contraceptives should add an additional barrier method as there is unknown whether lenvatinib may reduce the effectiveness of the hormonal contraceptives. All women who are of reproductive potential and who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.

    ** Sexual abstinence will be acceptable only when this is in line with the preferred and usual lifestyle of the subject.
18. Male subjects who are partners of women of childbearing potential must use or their partners must use a highly effective method of contraception (e.g., condom + spermicide, condom + diaphragm with spermicide, IUD) beginning at least 1 menstrual cycle prior to starting study drug(s), throughout the entire study period, and for 30 days after the last dose of study drug, unless they are sexually abstinent or have undergone a successful vasectomy. Those with partners using hormonal contraceptives must also be using an additional approved method of contraception, as described previously.
19. Voluntary provision of written informed consent and the willingness and ability to comply with all aspects of the protocol.

EXCLUSION CRITERIA

1. WHO Classification G3 neuroendocrine tumors of the pancreas and gastrointestinal tract.
2. Two or more prior lines of targeted agents-based therapy in pancreatic origin and any previous line of targeted therapy for gastrointestinal origin or any ongoing antiproliferative treatment for advanced/metastatic neuroendocrine tumors, with the exception of somatostatin analogues therapy.
3. More than one previous line of chemotherapy in pancreatic neuroendocrine tumors.
4. Previous chemotherapy in gastrointestinal neuroendocrine tumors.
5. Prior treatment with lenvatinib.
6. Subjects who have received any anti-cancer treatment within 21 days or any investigational agent within 30 days prior to the first dose of study drug and should have recovered from any toxicity related to previous anti-cancer treatment. This does not apply to the use of somatostatin analogues for symptomatic therapy.
7. Major surgery within 3 weeks prior to the first dose of study drug.
8. Subjects having > 1+ proteinuria on urine dipstick testing will undergo 24h urine collection for quantitative assessment of proteinuria. Subjects with urine protein ≥ 1 g/24h will be ineligible.
9. Gastrointestinal malabsorption, or any other condition in the opinion of the investigator that might affect the absorption of lenvatinib.
10. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina; myocardial infarction or stroke within 6 months prior to the first dose of study drug, or cardiac arrhythmia requiring medical treatment. The left ventricular ejection fraction in the echocardiogram must be of at least 50%.
11. Prolongation of QTcF interval to > 480 msec.
12. Bleeding or thrombotic disorders or use of anticoagulants, such as warfarin, or similar agents requiring therapeutic international normalized ration (INR) monitoring. Treatment with low molecular weight heparin (LMWH) is allowed.
13. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
14. Active infection (any infection requiring treatment).
15. Active malignancy within the past 5 years (except for definitely treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix).
16. Known intolerance or hypersensitivity to the active substance (or any of the excipients).
17. Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial.
18. Females who are pregnant or breastfeeding.
19. Documented active alcohol or drug abuse.
20. Patients with a prior history of non-compliance with medical regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Austria (2):
  - Universitätsklinik für Innere Medizin, Graz
  - Medizinische Universität Wien, Vienna
- Italy (8):
  - Spedali Civili di Brescia, Brescia
  - Instituto Oncologico Mediterraneo, Catania
  - Azienda Ospedaliero Universitaria Careggi - SC di Oncologia, Florence
  - IRST of Meldola, Meldola
  - Istituto Europeo di Oncologia - Unità di Oncologia Medica Gastrointestinale e Tumori Neuroendocrini, Milan
  - AOU Policlinico di Modena - DH Oncologico, Modena
  - IRCCS Napoli, Napoli
  - Hospital Universatorio de Verona, Verona
- Spain (10):
  - Hospital Virgen de la Victoria, Málaga, Andalusia
  - Hospital de Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Vall Hebrón, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Miguel Servet, Zaragoza
- United Kingdom (2):
  - Beatson Oncology Centre Gartnavel General Hospital, Glasgow
  - Christie Hospital, Manchester, Manchester

REFERENCES:
- [Derived] Ligero M, Hernando J, Delgado E, Garcia-Ruiz A, Merino-Casabiel X, Ibrahim T, Fazio N, Lopez C, Teule A, Valle JW, Tafuto S, Custodio A, Reed N, Raderer M, Grande E, Garcia-Carbonero R, Jimenez-Fonseca P, Garcia-Alvarez A, Escobar M, Casanovas O, Capdevila J, Perez-Lopez R. Radiomics and outcome prediction to antiangiogenic treatment in advanced gastroenteropancreatic neuroendocrine tumours: findings from the phase II TALENT trial. BJC Rep. 2023 Aug 2;1(1):9. doi: 10.1038/s44276-023-00010-0. PMID 39516643
- [Derived] Capdevila J, Fazio N, Lopez C, Teule A, Valle JW, Tafuto S, Custodio A, Reed N, Raderer M, Grande E, Garcia-Carbonero R, Jimenez-Fonseca P, Hernando J, Bongiovanni A, Spada F, Alonso V, Antonuzzo L, Spallanzani A, Berruti A, La Casta A, Sevilla I, Kump P, Giuffrida D, Merino X, Trejo L, Gajate P, Matos I, Lamarca A, Ibrahim T. Lenvatinib in Patients With Advanced Grade 1/2 Pancreatic and Gastrointestinal Neuroendocrine Tumors: Results of the Phase II TALENT Trial (GETNE1509). J Clin Oncol. 2021 Jul 10;39(20):2304-2312. doi: 10.1200/JCO.20.03368. Epub 2021 May 4. PMID 33945297

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment of patients was performed from 15/10/2015 until 08/09/2017 in participating hospitals.
Pre-assignment Details: A screening phase was designed with the purpose of stablishing protocol eligibility. Subjects who complete the baseline visit and continued to meet the criteria for inclusion/exclusion began the treatment phase of this study. A total of 123 patients were screened for enrolment into the study. 12 patients were screening failure. A total of 111 patients were included in the treatment phase of this study.
Groups:
- Neuroendocrine Tumors of the Pancreas: Patients with advanced/metastatic, histologically confirmed, grade 1/2 (G1/G2) of 2010 WHO (World Health Organization) classification neuroendocrine tumors of the pancreas after progression to a previous targeted agent.
  Treatment: Dosing schedule of 24 mg once a day of Lenvatinib (two 10-mg capsules + one 4-mg capsule)
  Lenvatinib
- Neuroendocrine Tumors of Gastrointestinal Tract: Patients with advanced/metastatic, histologically confirmed, grade 1/2 (G1/G2) of 2010 WHO (World Health Organization) classification neuroendocrine tumors of gastrointestinal tract after progression to somatostatin analogues Treatment: Dosing schedule of 24 mg once a day of Lenvatinib (two 10-mg capsules + one 4-mg capsule)
  Lenvatinib
Period: Overall Study
Arm/Group | Neuroendocrine Tumors of the Pancreas | Neuroendocrine Tumors of Gastrointestinal Tract
Started | 55 | 56
Completed | 28 | 28
Not Completed | 27 | 28
Not completed — Adverse Event | 11 | 14
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Sponsor discontinuation | 7 | 4
Not completed — Death | 1 | 1
Not completed — Other | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neuroendocrine Tumors of the Pancreas | Neuroendocrine Tumors of Gastrointestinal Tract | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.91 (10.36) | 61.48 (11.37) | 59.71 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 23 | 54
  Male | 24 | 33 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 54 | 56 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 3 | 3 | 6
  United Kingdom | 2 | 11 | 13
  Italy | 23 | 16 | 39
  Spain | 27 | 26 | 53
Menopausial Status [Count of Participants; unit: Participants] — Population: Only female patients are applicable to this category. Total females in cohort A (pancreatic tumor) are 31, however, for menopausal status, only information of 30 females is available. Information of menopausal status for 1 patient was not available.
  Participants
    number analyzed (Participants) | 30 | 23 | 53
    Premenopausal | 8 | 4 | 12
    Postmenopausal | 22 | 19 | 41
Time to Informed Consent (IC) signature [Mean (Standard Deviation); unit: years] — Population: This information was not available for some patients. It was only analysed when complete dates were provided.
  years
    number analyzed (Participants) | 38 | 44 | 82
    (all) | 4.95 (3.04) | 4.11 (3.9) | 4.5 (3.53)
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — ECOG Performance Scale is based in 5 grades:
  0.Fully active,able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    Grade 0 | 40 | 34 | 74
    Grade 1 | 15 | 22 | 37
Differentiation grade [Count of Participants; unit: Participants] — Differentiation grade is based in 2010 WHO Classification of neuroendocrine tumors according to Ki67 and mitotic count: patients must be Grade 1 or Grade 2 to be included in the trial. WHO Classification Grade 1 involves Ki67 ≤2% and mitotic count <2 mitoses x 10 HPF (High-Power Field); Grade 2 involves Ki67 3-20% and mitotic count 2-20 mitoses x 10 HPF (High-Power Field). Patients are assigned to a grade according to a histological diagnosis of the tumour (tissue biopsy analysis).
  Participants
    Grade 1 | 11 | 19 | 30
    Grade 2 | 40 | 33 | 73
    Not available | 4 | 4 | 8
Ki67 Expression [Mean (Standard Deviation); unit: Percent of cells with Ki67 Expression] — Population: This measure was not available for some participants.
  Percent of cells with Ki67 Expression
    number analyzed (Participants) | 54 | 54 | 108
    (all) | 9.57 (6.62) | 5.73 (4.91) | 7.65 (6.11)
Mitotic Count [Mean (Standard Deviation); unit: mitotic count] — mitotic count is defined as mitoses x 10 HPF (high powered field) Population: This measure was not available for some participants.
  mitotic count
    number analyzed (Participants) | 21 | 30 | 51
    (all) | 2.07 (2.01) | 4.25 (6.35) | 3.35 (5.11)
New York Heart Association (NYHA) classification [Count of Participants; unit: Participants] — Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    Class I | 11 | 8 | 19
    Class II | 1 | 0 | 1
    Class III | 0 | 0 | 0
    Class IV | 0 | 0 | 0
    Not applicable | 43 | 48 | 91
Diabetes [Count of Participants; unit: Participants]
  Yes | 21 | 4 | 25
  No | 31 | 47 | 78
  Not available | 3 | 5 | 8
Toxic Habits [Count of Participants; unit: Participants] — Documented drink of alcohol or smoke tobacco
  Participants
    Yes | 8 | 5 | 13
    No | 44 | 45 | 89
    Not available | 3 | 6 | 9
Hypertension [Count of Participants; unit: Participants]
  Yes | 22 | 30 | 52
  No | 30 | 21 | 51
  Not available | 3 | 5 | 8
Dyslipidaemia [Count of Participants; unit: Participants]
  Yes | 13 | 10 | 23
  No | 39 | 41 | 80
  Not available | 3 | 5 | 8
Kidney disease [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 51 | 51 | 102
  Not available | 3 | 5 | 8
Cardiovascular disease [Count of Participants; unit: Participants]
  Yes | 5 | 7 | 12
  No | 47 | 44 | 91
  Not available | 3 | 5 | 8
Operation for a primary tumor [Count of Participants; unit: Participants]
  Yes | 26 | 36 | 62
  No | 29 | 20 | 49
Operation for a metastatic tumor [Count of Participants; unit: Participants]
  Yes | 9 | 16 | 25
  No | 46 | 40 | 86
Functionality of tumor [Count of Participants; unit: Participants]
  Functional | 8 | 22 | 30
  Non-functional | 45 | 30 | 75
  Not available | 2 | 4 | 6
Origin of tumor [Count of Participants; unit: Participants] — Population: This category is only applicable to patients in Cohort B
  Participants
    number analyzed (Participants) | 0 | 56 | 56
    Ileum | 0 | 44 | 44
    Gastric | 0 | 1 | 1
    Colon | 0 | 3 | 3
    Rectum | 0 | 6 | 6
    Not available | 0 | 2 | 2
Tumor burden [Count of Participants; unit: Participants] — Tumor burden was assessed upon central radiology review, refers to the size of the tumor, and its reduction. So the tumor burden % refers to the decrease of the tumor size
  Participants
    reduction tumor burden <25% | 26 | 29 | 55
    reduction tumor burden 25-50% | 20 | 16 | 36
    reduction tumor burden >50% | 9 | 11 | 20
Previous Chemotherapy [Count of Participants; unit: Participants] — Population: This category is only applicable to patients in Cohort A.
  Participants
    number analyzed (Participants) | 55 | 0 | 55
    Yes | 18 | 0 | 18
    No | 37 | 0 | 37
Previous Chematherapy Treatment [Count of Participants; unit: Participants] — Population: This category is only applicable to patients in Cohort A that have previously received chemotherapy.
  Participants
    number analyzed (Participants) | 18 | 0 | 18
    Based on streptozotin | 5 | 0 | 5
    Based on Temozolomide | 8 | 0 | 8
    Other | 5 | 0 | 5
Previous anti-cancer agent with a targeted agent [Count of Participants; unit: Participants] — Population: This category is only applicable to patients in Cohort A.
  Participants
    number analyzed (Participants) | 55 | 0 | 55
    Yes | 55 | 0 | 55
    No | 0 | 0 | 0
Previous anti-cancer treatment with interferon [Count of Participants; unit: Participants] — Population: This category is only applicable to patients in Cohort B.
  Participants
    number analyzed (Participants) | 0 | 56 | 56
    Yes | 0 | 1 | 1
    No | 0 | 55 | 55
Previous anti-cancer treatment with somatostin analogues [Count of Participants; unit: Participants]
  Yes | 47 | 56 | 103
  No | 8 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Best Response Rate by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 Upon Central Radiologic Assessment
Description: Data cut-off for the primary study analysis will happen following after the last patient included in the study has performed the second tumor evaluation (week 18 after first dose of study drug as first evaluation will take place 6 weeks after first dose, following tumor assessment will take place every 12 weeks until documentation of disease progression or start of another anticancer therapy.
  Per Response Evaluation Criteria In Solid Tumors (RECIST v1.1) for target lesions: Complete Response (CR)= Disappearance of all target lesions; Partial Response (PR)= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; Progressive Disease (PD)=At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; Stable Disease (SD)= Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Overall Response (OR) = CR + PR.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroendocrine Tumors of the Pancreas | Neuroendocrine Tumors of Gastrointestinal Tract
Number analyzed (Participants) | 52 | 55
Participants
  Best Overall Response CR | 0 | 0
  Best Overall Response PR | 23 | 9
  Best Overall Response SD | 27 | 42
  Best Overall Response PD | 2 | 1
  Not evaluable | 0 | 3

2. Primary Outcome: Overall Response Rate (ORR) by RECIST v 1.1 Upon Central Radiologic Assessment
Description: Data cut-off for the primary study analysis will happen following after th e last patient included in the study has performed the second tumor evaluation (week 18 after first dose of study drug as first evaluation will take place 6 weeks after first dose, following tumor assessment will take place every 12 weeks until documentation of disease progression or start of another anticancer therapy
Time Frame: Up to 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | Neuroendocrine Tumors of the Pancreas | Neuroendocrine Tumors of Gastrointestinal Tract
Number analyzed (Participants) | 52 | 55
percentage of participants with response | 44.23 [30.73 to 58.58] | 16.36 [8.2 to 29.3]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from the date of treatment start (C1D1)to the date of first documentation of disease progression or death (whichever Occurs first) using RECIST 1.1. PFS censoring rules will follow FDA guidance in 2007
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroendocrine Tumors of the Pancreas | Neuroendocrine Tumors of Gastrointestinal Tract
Number analyzed (Participants) | 55 | 56
Participants
  No PD/ No Exitus | 12 | 12
  PD | 34 | 36
  Exitus (No PD) | 5 | 7
  Not available | 4 | 1

4. Secondary Outcome: Number of Participants With Early Tumor Shrinkage (ETS)
Description: To calculate early tumor shrinkage (ETS) rate, patients were classified as responders/non-responders after a period of 6 weeks (first post-baseline tumor assessment). Those who achieved a 20% reduction in target lesions after the first 6 weeks of treatment were classified as responders.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroendocrine Tumors of the Pancreas | Neuroendocrine Tumors of Gastrointestinal Tract
Number analyzed (Participants) | 52 | 51
Participants
  Non-responders | 32 | 46
  Responders | 20 | 5

5. Secondary Outcome: Deepness of Response (DpR)
Description: (DpR) defined as percentage of maximum tumor shrinkage observed at the nadir compared with baseline
Time Frame: Up to 18 months
Measure: Median (Inter-Quartile Range); unit: Percentage of tumour reduction
Arm/Group | Neuroendocrine Tumors of the Pancreas | Neuroendocrine Tumors of Gastrointestinal Tract
Number analyzed (Participants) | 52 | 56
Percentage of tumour reduction | -26.28 [-39.86 to -16.13] | -15.34 [-26.14 to -6.67]

6. Secondary Outcome: Tumour Shrinkage
Description: Number of patients that exhibited a deepness of response lower than 0%.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroendocrine Tumors of the Pancreas | Neuroendocrine Tumors of Gastrointestinal Tract
Number analyzed (Participants) | 52 | 52
Participants
  No tumor shrinkage | 6 | 6
  Tumor shrinkage | 46 | 46

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Neuroendocrine Tumors of the Pancreas | Neuroendocrine Tumors of Gastrointestinal Tract
All-Cause Mortality (participants affected / at risk) | 21/55 | 29/56
Serious Adverse Events (participants affected / at risk) | 23/55 | 24/56
Other Adverse Events (participants affected / at risk) | 55/55 | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neuroendocrine Tumors of the Pancreas (N=55) | Neuroendocrine Tumors of Gastrointestinal Tract (N=56)
Abdominal Pain (Gastrointestinal disorders) | 3 | 3
Intestinal Obstruction (Gastrointestinal disorders) | 3 | 3
Acute Kidney Injury (Renal and urinary disorders) | 2 | 2
Anal Abscess (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Benign Neoplasm of bladder (Renal and urinary disorders) | 1 | 0
Bile duct steneosis (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Choleocistitis (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Colon Operation (Gastrointestinal disorders) | 1 | 0
Confusional state (Nervous system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic stroke (Cardiac disorders) | 1 | 0
Hepatic infection (Infections and infestations) | 1 | 0
Hyperamylaseamia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Lower Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pancratitis acute (Gastrointestinal disorders) | 1 | 0
Abdominal Abcess (Gastrointestinal disorders) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Blood bilirubin increased (Hepatobiliary disorders) | 0 | 1
Choleolithiasis (Hepatobiliary disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastroduodenal haemmorhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 1
Gatrointestinal Toxicity (Gastrointestinal disorders) | 0 | 1
General Physical Health detereoration (General disorders) | 0 | 1
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Kidney infection (Renal and urinary disorders) | 0 | 1
Lymphoedema (Blood and lymphatic system disorders) | 0 | 1
Metastases to large intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myocardial infactation (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Pyrexia (Infections and infestations) | 0 | 1
Rectal Haemmorhage (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Small Intestin perforation (Gastrointestinal disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuroendocrine Tumors of the Pancreas (N=55) | Neuroendocrine Tumors of Gastrointestinal Tract (N=56)
Abdominal pain (Gastrointestinal disorders) | 55 (1428) | 56 (1220)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT02678780/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT02678780/SAP_001.pdf